CLINICAL TRIAL: NCT00914160
Title: A Relative Bioavailability Study of Diclofenac Sodium 50 mg Enteric-Coated Tablets Under Non-Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Diclofenac Sodium 50 mg Enteric-Coated Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B-08133
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-06

CONDITIONS: Inflammation
Keywords: Anti-inflammatory
MeSH Terms: conditions — Inflammation | interventions — Diclofenac

ARMS (3):
- 1 (Experimental): Diclofenac Sodium 50 mg Tablets Under Fasting Conditions (Geneva Pharmaceuticals, Inc)
  Interventions: Drug: Diclofenac Sodium 50 mg Tablets Under Fasting Conditions (Geneva Pharmaceuticals, Inc)
- 2 (Experimental): Diclofenac Sodium 50 mg Tablets Under Fed Conditions (Geneva Pharmaceuticals, Inc)
  Interventions: Drug: Diclofenac Sodium 50 mg Tablets Under Fed Conditions (Geneva Pharmaceuticals, Inc)
- 3 (Active Comparator): Voltaren 50 mg Tablets Under Fed Conditions (Geigy Pharmaceuticals)
  Interventions: Drug: Voltaren 50 mg Tablets Under Fed Conditions (Geigy Pharmaceuticals)

INTERVENTIONS:
Drug: Diclofenac Sodium 50 mg Tablets Under Fasting Conditions (Geneva Pharmaceuticals, Inc)
  Arms: 1
Drug: Diclofenac Sodium 50 mg Tablets Under Fed Conditions (Geneva Pharmaceuticals, Inc)
  Arms: 2
Drug: Voltaren 50 mg Tablets Under Fed Conditions (Geigy Pharmaceuticals)
  Arms: 3

SUMMARY:
To demonstrate the relative bioavailability of Diclofenac Sodium 50 mg enteric-coated tablets under non-fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 1993-08; Primary Completion 1993-09 (Actual); Study Completion 1993-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul D. Larsen, M.D., Principal Investigator — Red River Clinic